CLINICAL TRIAL: NCT05257759
Title: Use of Neurostimulation As a Tool for Reconditioning the Neuromuscular System of Patients Admitted to the ICU for Septic Shock: a Single-center Randomized Pilot Study
Brief Title: Use of Neurostimulation As a Tool for Reconditioning the Neuromuscular System of Patients Admitted to the ICU for Septic Shock
Acronym: STIMUREA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment for the study
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANDREU AOI 2021
Record Dates: First submitted 2022-01-25; First posted 2022-02-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Septic Shock
Keywords: reanimation neuromyopathy
MeSH Terms: conditions — Shock, Septic | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard support (Active Comparator)
  Interventions: Other: Usual care; Other: Evaluation of the neuromuscular system
- Standard treatment coupled with electro-stimulation sessions (Experimental)
  Interventions: Other: Usual care; Other: Electrostimulation; Other: Evaluation of the neuromuscular system

INTERVENTIONS:
Other: Usual care — Standard management offered in the intensive care unit
Other: Electrostimulation — The patients included will receive throughout their stay, in addition to the standard care offered in the department, electrical nerve stimulation. The ES will be applied to the tibial nerve to allow contraction of the plantar flexors. The protocol will be applied twice a day, 5-7 days a week and will have the following characteristics: stimulation frequency 100Hz, pulse width 1ms, intensity allowing the development of 5-10% of the maximum tetanic force obtained during the force-frequency relation, contraction time 20s, recovery time 20s, for a total of 25 contractions per session.
  Arms: Standard treatment coupled with electro-stimulation sessions
Other: Evaluation of the neuromuscular system — Will be performed within 48 hours of admission to the ICU and at D7 of admission.
  Includes:
  * electrical stimulations (at an intensity to obtain 10% of the maximum M wave) in the leg at different frequencies with recording of the force developed by force sensor
  * maximum and submaximal electrical stimulation of the leg with recording of the electrophysiological response by surface electrodes applied to the leg muscles, to evaluate muscular and spinal excitability.
  * MRC scale to assess the motor function of different muscle groups of the lower and upper of the lower and upper limbs, depending on the patient's clinical condition.
  * Maximum Voluntary Contractions (MVC) to evaluate the muscular strength of the plantar flexors, depending on the patient's clinical condition.

SUMMARY:
Patients hospitalized in the ICU are likely to develop sarcopenia due to a progressive and generalized decrease in muscle mass that is responsible for generalized muscle weakness known as resuscitation neuromyopathy. This neuromyopathy is known make weaning from mechanical ventilation more difficult, which prolongs the hospitalization of patients in the ICU and in hospital. The factors identified as being partly responsible for this neuromyopathy are: immobilization, undernutrition, prolonged duration of mechanical ventilation, inflammation (notably secondary to sepsis), and multivisceral failure. These factors are essentially found in patients in septic shock, which represents about 20% of patients admitted to the ICU, with a mortality rate close to 50%. If the management of septic shock is now well codified (i.e. vascular filling, antibiotics and/or treatment of the infectious focus by surgery +/- organ replacement therapy) as well as the early rehabilitation of ICU patients, no treatments has yet been proven to be effective in limiting the appearance of resuscitation neuromyopathy. For the last ten years, research using electrostimulation (ES) to improve muscle contraction seems to give encouraging results, both for length of hospital stay and the duration of mechanical ventilation, notably through the preservation or a significant increase in muscle strength. On the other hand, other studies did not show a significant effect on muscle strength. These conflicting results are partly related to the heterogeneity of the populations included in the studies and to the different ES approaches used to assess and recondition motor function.

In the present STIMUREA study, an original approach is proposed based on experimental research work carried out for many years within U1093 (Pr Charalambos Papaxanthis) which focuses on ES, not of the muscle surface as in most studies carried out in the ICU, but an approach based on ES of the motor nerve. Indeed, the intensity of ES used in previous studies was based on a maximum tolerated intensity leading to a direct recruitment of the most fatiguable motor units (via the activation of motor axons) but leading, in fine, to a decrease in muscle strength. The U1093 research team and previous studies have shown that protocols using high stimulation frequencies (100Hz) associated with pulse widths of 1ms and delivered at low intensities (5-10% of the maximum voluntary contraction, MVC) at the level of the motor nerve, could increase the force developed during the contraction, while decreasing the discomfort induced by the high intensities. This increase in force would be due to the indirect activation of motor neurons via large diameter sensory afferents, thus leading to a recruitment of motor units similar to that observed during voluntary contractions. In a very recent study conducted in our laboratory (INSERM U1093), it was demonstrated that the application of ES to the motor nerve at low intensities did not induce discomfort in healthy subjects, but could induce substantial strength gains (+25%) with adaptations occurring at both in the muscles and the nerves.

The proposed study is an innovative, randomized, pilot study based on motor nerve ES in a highly selected population of ICU patients in septic shock and therefore with a high risk of developing neuromyopathy, which is responsible for a significant increase in morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to the ICU for :

  * Sepsis as defined by the presence of an infection, of known or suspected origin + organ dysfunction with a SOFA score ≥ 2
  * Or septic shock defined by sepsis with persistent hypotension requiring vasopressors to maintain mean artérial blood pressure ≥ 65 mmHg and serum lactate level > 2 mmol/l despite adequate vascular filling
* After obtaining informed consent from a relative/trusted person or patient included in an emergency situation
* Patient affiliated to national health insurance.

Exclusion Criteria:

* Patient with a contraindication to the application of ES (e.g. pacemaker, defibrillator)
* Patient with a diagnosis of deep vein thrombosis and/or pulmonary embolism, confirmed and treated within the last 48 hours
* Patient with cardiac arrest prior to study inclusion
* Patient for whom a decision to limit or stop treatment has been made by the medical team
* Patients with a very poor prognosis in the very short term due to major co-morbidities (Child Pugh score C cirrhosis, terminal cancer, neuro-evolutionary disease with no treatment plan...)
* Patients with known neuro-orthopaedic and sensory disorders prior to inclusion, whether of originating in the spinal cord, nerve or brain.
* Person subject to a legal protection measure (curatorship, guardianship)
* Pregnant, parturient or breastfeeding women.

Secondary Exclusion Criteria:

- Patients receiving curare therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
change of the muscle force in newton meters (Nm) of the plantar flexors in response to electrical stimulation of the tibial nerve | Between inclusion and Day 7 of admission in the intensive care unit
  change of muscle strength between inclusion and at Day 7 (between Day 7 and Day 8) of admission in the intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No